CLINICAL TRIAL: NCT05092230
Title: Frequency of Pompe Disease in Patients Followed at CERCA for Myalgia With or Without Hyper Ckemia
Brief Title: Frequency of Pompe Disease in Patients With Myalgia With or Without Hyper Ckemia - Data From the Reference Center (CERCA)
Acronym: POEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: POEM
Record Dates: First submitted 2021-08-23; First posted 2021-10-25 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Pompe Disease
Keywords: frequency,; MARTINIQUE; observational study; myalgia; reference center for rare diseases
MeSH Terms: conditions — Glycogen Storage Disease Type II; Myalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pompe's disease is a lysosomal storage disease of autosomal recessive genetic transmission due to a deficiency in acid alpha glucosidase. This enzyme deficiency leads to glycogen overload in all cells but with a more marked expression in muscle cells. There is a great variability in the clinical manifestations and in the age of onset of symptoms depending on whether the enzyme deficiency is partial or total. The prevalence is estimated at 1 in 40,000. There is a specific treatment based on enzyme replacement therapy

DETAILED DESCRIPTION:
Patients include: clinical examination, enzyme activity assay, muscle testing, cardiological and respiratory workup. Lowered enzyme activity suggests a pathogenic genetic variant to be identified. The secondary objective is to propose genetic counselling and a family investigation in order to identify relatives who are also affected.

ELIGIBILITY:
Inclusion Criteria:

* • both sexes

  * with permanent myalgia, spontaneous or on effort,
  * with or without muscle deficit,
  * with or without HyperCkemia
  * without known etiologies
  * Age from 6 to 80 years
  * consulting for the first time or followed at CERCA
  * giving their free and informed consent to participate after information on the research
  * Affiliated to the social security system

Exclusion Criteria:

* Person placed under guardianship and/or curatorship
* Myalgias related to a known etiology

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient 6 to 80 years of age or consulting for the first time or followed at CERCA Martinique with permanent myalgia, spontaneous or on effort,
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure | The recruitment will take place in our specialized center for the management and follow-up of patients with neuromuscular pathology. A total of 100 patients are likely to be included in the study during the years 2020-2022
  To estimate the frequency of Pompe's disease in men and women with permanent, spontaneous or exertional myalgia consulting for the first time or followed in our center. This criterion will be evaluated by biochemical and genetic analyses. Improvement of diagnostic deficiency and genetic counseling is envisaged. A discussion could be opened for these patients regarding the application of enzyme replacement therapy.

SECONDARY OUTCOMES:
Muscle testing | 2 years
  - Muscle Testing using Medical Research Counsil scale (MRC scale, total score ranging from 0 to 5)
Cardiological check-up | 2 years
  - ECG : QRS Complex and short PR space (milliseconde)
Respiratory check-up | 2 years
  - Chest radiography (non mesurable)
Genetic counselling activity | 2 years
  - Genetic counseling appointment (non mesurable)
Muscle testing | 2 years
  - 6-minute walk test (number of metres in 6 minutes)
Muscle testing | 2 years
  motor function scale (french " MFM ") (32 items rated on a 4-point Likert scale)
Muscle testing | 2 years
  ElectroNeuroMyogram (ENMG) with measurement of nerve conduction velocities (m/s)
Cardiological check-up | 2 years
  - Holter-ECG during 24h : heart rhythm abnormality (beat per minute)
Cardiological check-up | 2 years
  Measurement of Brain Natriuretic Peptid (BNP) (ng/L)

OTHER OUTCOMES:
Respiratory check-up | 2 years
  - Blood gas : Pa O2 (mmHg) Pa CO2 (mmHg), pH
Respiratory check-up | 2 years
  Maximum Expiratory Volume in the 1st second during forced expiration, "VEMS"(L)
Respiratory check-up | 2 years
  o Functional Vital Capacity, " CV " (L)
Respiratory check-up | 2 years
  o percentage of FEV1 to vital capacity "VEMS%CV"
Respiratory check-up | 2 years
  o Mean Expiratory Flow " DEM) (L/s)
Respiratory check-up | 2 years
  - Polysomnography : index number of apneas per hour
Genetic counselling activity | 2 years
  - Biological sampling of relatives (non mesurable)
Cardiological check-up | 2 years
  echocardiogram (FEVG, measurement of cardiac walls in mm)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lukacs Z, Nieves Cobos P, Wenninger S, Willis TA, Guglieri M, Roberts M, Quinlivan R, Hilton-Jones D, Evangelista T, Zierz S, Schlotter-Weigel B, Walter MC, Reilich P, Klopstock T, Deschauer M, Straub V, Muller-Felber W, Schoser B. Prevalence of Pompe disease in 3,076 patients with hyperCKemia and limb-girdle muscular weakness. Neurology. 2016 Jul 19;87(3):295-8. doi: 10.1212/WNL.0000000000002758. Epub 2016 May 11. PMID 27170567
- [Background] Taisne N, Desnuelle C, Juntas Morales R, Ferrer Monasterio X, Sacconi S, Duval F, Sole G, Flipo RM, Lacour A, Vermersch P, Cardon T. Bent spine syndrome as the initial symptom of late-onset Pompe disease. Muscle Nerve. 2017 Jul;56(1):167-170. doi: 10.1002/mus.25478. Epub 2016 Nov 30. PMID 27862019